CLINICAL TRIAL: NCT04427475
Title: Study on the Prediction of Immunotherapeutic Effect of Advanced Non-small Cell Lung Cancer by Detection of Plasma Exosomes
Brief Title: Prediction of Immunotherapeutic Effect of Advanced Non-small Cell Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jialei Wang, Principal Investigator, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MIRNA-SEP-01
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: NSCLC Patients

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pabolizumab (Other): Baseline plasma samples were collected before the treatment, and the efficacy was evaluated once every two treatment cycles.
  Interventions: Drug: pabolizumab
- nafulizumab (Other): Baseline plasma samples were collected before the treatment, and the efficacy was evaluated once every two treatment cycles.
  Interventions: Drug: nafulizumab

INTERVENTIONS:
Drug: pabolizumab — 100 patients with stage IV EGFR / ALK wild-type NSCLC (squamous cell carcinoma patients do not need to be detected) who received anti-PD-1 (pabolizumab) treatment combined with chemotherapy as the first-line treatment were enrolled in the center. Baseline plasma samples were collected before the treatment, and the efficacy was evaluated once every two treatment cycles. At the same time, plasma samples were collected at key nodes until the patient's progress.
  Arms: pabolizumab
Drug: nafulizumab — nafulizumab
  Arms: nafulizumab

SUMMARY:
To detect the difference of PD-L1 and miRNA expression profiles of exosomes in NSCLC patients before and after immunotherapy, and to explore the potential of plasma exosomes PD-L1 and miRNAs as biomarkers to predict the therapeutic effect of NSCLC on anti-PD-1 / PD-L1.

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent.
2. The age is greater than or equal to 18 years old.
3. There is at least one measurable focus according to the RECIST 1.1 standard
4. EGFR / ALK detection is not needed in patients with metastatic (stage IV) EGFR / ALK wild-type NSCLC confirmed by histology or cytology and in patients with squamous cell carcinoma.
5. Cohort 1: patients receiving anti-PD-1 (pabolizumab) treatment combined with chemotherapy as the first-line treatment Cohort 2: patients who received the second-line treatment of anti-PD-1 single drug (nafulizumab) for the progress of disease after chemotherapy with platinum containing dual drugs
6. ECoG score is 0, 1 or 2.
7. No serious blood system, heart, lung, liver and kidney dysfunction and immune deficiency.
8. Hemoglobin (HB) ≥ 9g / dl; leukocyte (WBC) ≥ 3 * 109 / L; neutrophil (ANC) ≥ 1.5 * 109 / L; platelet (PLT) ≥ 75 * 109 / L.
9. Men or women of childbearing age are willing to take contraceptive measures in the experiment.
10. Estimated survival time ≥ 3 months.

Exclusion Criteria:

1. Histologically, small cell and non-small cell mixed lung cancer.
2. Pregnant or nursing women.
3. Any unresponsive > CTCAE Level 2 toxicity caused by past anti-tumor treatment
4. Serum creatinine clearance < 30 ml / min (calculated by Cockcroft Gault formula)
5. Liver dysfunction, defined as:

   1. Serum (total) bilirubin > 1.5 × upper limit of normal value (ULN)
   2. Serum AST / SGOT or ALT / SGPT > 2.5 × ULN (liver metastasis > 5 × ULN)
   3. Alkaline phosphatase level > 2.5 × ULN (liver metastasis > 5 × ULN, or bone) at baseline Transfer patients > 10 × ULN)
6. Have a history of uncontrollable or symptomatic angina, arrhythmia or congestive heart failure.
7. Symptomatic brain metastasis or meningeal metastasis.
8. In the past 5 years, she has had or is suffering from other histological types of malignant tumors, except for cervical carcinoma in situ and fully treated skin basal cell carcinoma or squamous cell carcinoma.
9. Have active, or have had and may recur autoimmune diseases. However, subjects with type I diabetes, hypothyroidism requiring hormone replacement therapy only, skin diseases without systemic treatment (such as vitiligo, psoriasis or alopecia), or no relapse without external triggers are expected.
10. Diagnosis of immunodeficiency or systemic hormone therapy (e.g., hormone therapy equivalent to > 10 mg prednisone per day) or any other form of immunosuppressive therapy within 7 days before the first administration.
11. Patients with known history of human immunodeficiency virus (HIV) infection and / or acquired immunodeficiency syndrome. Subjects with active hepatitis B or active hepatitis C
12. Grade 2 pneumonia caused by radiotherapy and chemotherapy (grade 2 pneumonia without systemic hormone treatment recovers to grade 1 or below within 14 days, if the researcher judges that there is no risk of recurrence, it can be included in the group for screening).
13. Have interstitial lung disease and the disease has symptoms.
14. During the study period, radiotherapy is planned for the target focus.
15. Plan to use other anti-tumor therapy during the study period.
16. Patients with serious or uncontrolled systemic diseases who are not suitable for the study or may affect the compliance of the other party's case. Subjects' complications or other conditions may affect compliance with the protocol or may not be suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
PD-L1 expression profiles of exosomes | through study completion, an average of 1 year
  detect the difference of PD-L1 expression profiles of exosomes in NSCLC patients before and after immunotherapy
miRNA expression profiles of exosomes | through study completion, an average of 1 year
  detect the difference of miRNA expression profiles of exosomes in NSCLC patients before and after immunotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer hospital Fudan University, Shanghai, Shanghai Municipality, China